CLINICAL TRIAL: NCT05698160
Title: Biomarkers and Prediction of Tigecycline Induced Coagulation Dysfunction Based on Multi-omics and Machine Learning Techbology
Brief Title: Biomarkers and Prediction of Tigecycline Induced Coagulation Dysfunction
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-LCYJ-PY-14
Record Dates: First submitted 2023-01-16; First posted 2023-01-26 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-01

CONDITIONS: Blood Coagulation Disorder
Keywords: Tigecycline; Blood Coagulation Disorder; multi-omics; machine learning techbology
MeSH Terms: conditions — Blood Coagulation Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- coagulation dysfunction group: The critically ill patients in intensive care unit showed coagulation dysfunction after treated with tigecycline.
- non-coagulation dysfunction group: The critically ill patients in intensive care unit showed normal coagulation function after treated with tigecycline.

SUMMARY:
This study is to screen out the biomarkers and establish the model to predict coagulation dysfunction induced tigecycline

DETAILED DESCRIPTION:
The critically ill patients treated with tigecycline in in tensive care unit will be recruited and divided into tigecycline-induced coagulation dysfunction group and non-coagulation dysfunction group. The multi-omics will be used to screen out biomarkers for early prediction of coagulation dysfunction caused by tigecycline. Afterwards, machine learning methods will be adopted to establish the the early prediction model of tigecycline-induced coagulation dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients receiving tigecycline treatment in the Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
* Intravenous tigecycline ≥ 3 days
* Monitoring the plasma concentration of tigecycline

Exclusion Criteria:

* Missing clinical data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The critically ill patients treated with tigecycline in the Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Biomarkers associated with the coagulation dysfunction induced tigecycline | January 2023-December 2025
  Multi-omics will be adopted to screen out biomarkers associated with the coagulation dysfunction induced by tigecycline.

SECONDARY OUTCOMES:
Prediction model for coagulation dysfunction induced by tigecycline | January 2023-December 2025
  Machine learning techbology will be adopted to establish the prediction model for coagulation dysfunction induced by tigecycline